CLINICAL TRIAL: NCT02810535
Title: Local IgE in Subjects With Allergic or Non-allergic Rhinitis
Acronym: LISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Zielen, Professor of pediatrics, allergy, pneumology, cystic fibrosis, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FRA.LISA.2015
Record Dates: First submitted 2016-05-31; First posted 2016-06-23 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Perennial Rhinitis
Keywords: Local IgE; Non-allergic rhinitis; Allergic rhinitis to house dust mite
MeSH Terms: conditions — Common Cold | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Allergic rhinitis (Active Comparator): Clinical observation of 24 subjects with nasal symptoms and positive prick test for house dust mite
  Interventions: Other: Observation
- Non-allergic rhinitis (Experimental): Clinical observation of 24 subjects with nasal symptoms and negative prick test for house dust mite
  Interventions: Other: Observation
- Healthy Control (Other): Clinical observation of 20 subjects without nasal symptoms and with negative prick test
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Visit 1:
  * Physical examination (inspection of nasopharynx, auscultation of heart and lungs)
  * Completion of a Health Questionnaire
  * Lung function testing with spirometry
  * Skin prick test
  Visit 2:
  * Physical examination (inspection of nasopharynx, auscultation of heart and lungs)
  * Measurement of nitric oxide in expired air (FeNO)
  * Taking nasal secretion samples with a cotton carrier for 15 min
  * Nasal provocation test with dust mite
  * Blood sample collection to define blood count, IgE and specific IgE

SUMMARY:
The purpose of the study is to investigate the incidence of non-allergic rhinitis on a not selected group of young students (n=100-300). Students will be selected by public posting. In all students an allergy skin test will be performed. Then the local IgE of 24 subjects with non-allergic rhinitis will be compared to the local IgE of 24 subjects with allergic rhinitis and positive prick test to house dust mite. In addition 20 controlls will be investigated. Based on these investigations, the importance of local IgE and the IgE spectrum in conjunction with rhinitis should be further clarified.

DETAILED DESCRIPTION:
20% of Germans suffer from seasonal or all-season rhinitis. Despite typical allergic symptoms, in a part of the affected patients (about 10-20%) an allergy cannot be found on skin prick test or blood. Therefore, the planned trial will investigate the incidence of allergic and non-allergic rhinitis in a non selected group of young students (n=100-300). The hypothesis postulates that in test subjects with non-allergic rhinitis the allergy can only be proven locally in nasal secretion.

From the initial large cohort of patients, 24 subjects with house dust mite allergy and allergic rhinitis and 24 patients with non-allergic rhinitis will be selected and investigated in more detail at a second visit. At the second visit, blood and nasal secretion (measurement of local IgE) will be taken from all pre-selected 48 patients. At visit 2 a nasal provocation test with house dust mite allergen will be performed in all patients to compare nasal symptoms with the results of local IgE between patient groups. In addition the same investigations will be performed in a group of 20 healthy non-allergic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Seasonal or all-season symptoms of an allergic or non-allergic rhinitis
* Healthy non-allergic subjects

Exclusion Criteria:

* Patients: Age <18 and > 45
* Other severe diseases (e.g. Cystic fibrosis, diseases with immunosuppression, malignant diseases)
* Previously occurred allergic shock
* Pregnancy and lactation
* Participation in another clinical trial within the last 30 days
* Inability to measure the length and the consequences of the study
* Frequent use of medication which could not be discontinued in the defined time before enrollment: nasal vasoconstrictors 1 day; antihistamines 3 days; nasal steroids 7 days; oral cortison 4 weeks; leukotriene antagonists and cromolyn 2 days before NPT

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Comparison of IgE between 24 subjects with non-allergic rhinitis, 24 subjects with allergic rhinitis and 20 healthy subjects. | one year

SECONDARY OUTCOMES:
Comparison of specific IgE between 24 subjects with non-allergic rhinitis, 24 subjects with allergic rhinitis and 20 healthy subjects. | one year
Correlation between Peak Nasal Inspiratory Flow as well as the nasal symptoms in nasal provocation test and local specific IgE. | one year
Explorative Measures: Comparison of the nasal and serum epitope spectrum with the new mite specific IgE component-chip in subjects with allergic rhinitis. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Professor, Principal Investigator — Department for children and adolescents, division of allergy, pneumology, and cystic fibrosis
Locations (1):
- Goethe University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bez C, Schubert R, Kopp M, Ersfeld Y, Rosewich M, Kuehr J, Kamin W, Berg AV, Wahu U, Zielen S. Effect of anti-immunoglobulin E on nasal inflammation in patients with seasonal allergic rhinoconjunctivitis. Clin Exp Allergy. 2004 Jul;34(7):1079-85. doi: 10.1111/j.1365-2222.2004.01998.x. PMID 15248853
- [Background] Litvyakova LI, Baraniuk JN. Nasal provocation testing: a review. Ann Allergy Asthma Immunol. 2001 Apr;86(4):355-64; quiz 364-5, 386. doi: 10.1016/S1081-1206(10)62478-7. PMID 11345277
- [Result] Buslau A, Voss S, Herrmann E, Schubert R, Zielen S, Schulze J. Can we predict allergen-induced asthma in patients with allergic rhinitis? Clin Exp Allergy. 2014 Dec;44(12):1494-502. doi: 10.1111/cea.12427. PMID 25270425
- [Result] Campo P, Rondon C, Gould HJ, Barrionuevo E, Gevaert P, Blanca M. Local IgE in non-allergic rhinitis. Clin Exp Allergy. 2015 May;45(5):872-881. doi: 10.1111/cea.12476. PMID 25495772
- [Result] Huggins KG, Brostoff J. Local production of specific IgE antibodies in allergic-rhinitis patients with negative skin tests. Lancet. 1975 Jul 26;2(7926):148-50. doi: 10.1016/s0140-6736(75)90056-2. PMID 49744
- [Derived] Eckrich J, Hinkel J, Fischl A, Herrmann E, Holtappels G, Bachert C, Zielen S. Nasal IgE in subjects with allergic and non-allergic rhinitis. World Allergy Organ J. 2020 Jun 23;13(6):100129. doi: 10.1016/j.waojou.2020.100129. eCollection 2020 Jun. PMID 32612737